CLINICAL TRIAL: NCT04518774
Title: The Safety Assessment of Ex-Vivo Expanded Allogeneic γδT Cells in Hepatocellular Carcinoma Patients in Phase 1 Clinical Trial
Brief Title: Allogeneic "Gammadelta T Cells (γδ T Cells)" Cell Immunotherapy in Phase 1 Hepatocellular Carcinoma Clinical Trial
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Beijing GD Initiative Cell Therapy Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JDH-HCC-002
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: allogeneic γδT cells; hepatocellular carcinoma; adoptive immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic γδT cell immunotherapy (Experimental): Patients will receive 3 cycles of ex-vivo expanded allogeneic γδT cells treatments, at four-weeks' intervals, each cycle has 2 infusions. Ex-vivo expanded γδT cells are transfused to patients in a dosage escalated manner (Dose escalation, 1×107, 3×107, 9×107 per kg of body weight).
  Interventions: Biological: Ex-vivo expanded allogeneic γδT cells

INTERVENTIONS:
Biological: Ex-vivo expanded allogeneic γδT cells — Cells will be extracted from a healthy donor by apheresis, followed by ex-vivo expansion and activation. The ex-vivo expanded γδT cells from donors will be adoptively transfused.

SUMMARY:
This study aims to evaluate the safety, tolerability and efficacy of ex-vivo expanded allogeneic γδT cells obtained from a blood-related donor of hepatocellular carcinoma patients.

DETAILED DESCRIPTION:
This study is a single-center, non-randomized, open label, no control, prospective clinical trial to evaluate the safety, tolerability and efficacy of ex-vivo expanded allogeneic γδT cells from of a blood-related donor of Hepatocellular Carcinoma (HCC) Patients. This study will include the following sequential phases: sign informed consent, γδT cell pre-culture, screening and registration to the trial, apheresis, γδT cell preparation, treatments and follow-ups.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Patients should sign informed consent form voluntarily before the trail and comply with the requirements of this study.
2. Age 18 years up to the age of 65 (≤65), gender unlimited.
3. Hepatocellular Carcinoma diagnosed according to the 2018 edition of the EASL guidelines. Patients should accept liver biopsy voluntarily and histopathologically diagnosed with HCC.
4. Interventional therapy (e.g. TACE), RFA or radiation therapy should be at least 2 weeks prior to γδT cell transfusion; surgical treatment should be at least 1 month prior to γδT cell transfusion. Patients can take the first- or second-line targeted drugs recommended by the guidelines, such as lenvatinib or sorafenib.
5. Liver function: Child-Pugh class A/B (5-9)
6. Eastern Cooperative Oncology Group (ECOG) Performance score≤2.
7. Life expectancy of at least 1 year.
8. Patients combined with HBV infection require antiviral treatment with nucleoside analogues; patients combined with HCV infection require direct-acting antiviral agent (DAA) treatment.
9. Male and female patients of reproductive potential must agree to use birth control during the study and for at least 30 days post study.

Patient Exclusion Criteria:

1. Patients combined with HAV, HEV, HIV or other infectious diseases.
2. Acute infections, gastrointestinal bleeding, etc. occurred within 30 days before screening.
3. Women who are pregnant (urine/blood pregnancy test positive) or lactating; patients with severe autoimmune diseases; patients with uncontrolled infectious diseases.
4. Major organs dysfunction:

   * Peripheral blood: WBC<1.0×109/L, PLT <60×109/L, Hb <86g/L;
   * Coagulation: INR>2.3, PT>18s;
   * Liver function: ALB<28g/L, TBIL>51mmol/L, ALT/AST>5 times the upper limit of normal, CREA>1.5 times the upper limit of normal.
5. Combined with other severe organic diseases or mental illnesses, including any uncontrolled clinically significant systematic diseases such as urinary, circulatory, respiratory, neurological, psychiatric, digestive, endocrine and immune diseases.
6. Allergic constitution, history of allergies to blood products, known to be allergic to test substances.
7. Immunosuppressive or systemic cytotoxic drugs may require within 6 months prior to screening or during the study; 6 months prior to screening accepted other cell therapies including NK, CIK, DC, CTL and stem cell therapy etc.; immunotherapy such as PD-1 and PD-L1 antibodies.
8. Patients currently participating in other clinical trials who may violate this treatment plan and observations.
9. Those who are unable or unwilling to provide informed consent or who are unable to comply with the research requirements.
10. Any situation that investigators believe the risk of the subjects is increased or results of the trial are disturbed: patients with any serious acute or chronic physical or mental illness, or laboratory abnormalities.

Donor Inclusion Criteria:

1. Sign informed consent form.
2. Age 18 years up to the age of 50 (≤50), gender unlimited.
3. Relative to patients (unrestricted to blood relationship).
4. Apheresis available.
5. PLT≥100×109/L with normal APTT or PT.

Donor Exclusion Criteria:

1. History of any severe clinical diseases or other severe organic diseases, including any history of clinically significant systematic diseases such as cardiovascular, urinary, circulatory, respiratory, neurological, psychiatric, digestive and endocrine diseases. History of high blood pressure or systolic pressure>140 mmHg, diastolic pressure>90 mmHg in screening stage. Any situation that investigators believe is clinically significant or with other severe diseases unsuitable of apheresis.
2. Arterial thrombosis or venous thrombosis history 12 months prior to the trial or hemorrhagic tendency or history 2 months prior to the trial; oral administration of anticoagulation drugs (e. g. aspirin and warfarin).
3. Active or history of autoimmune diseases including but not restricted to SLE, psoriasis, RA, IBD and HT. Apart from hypothyrosis which can be controlled by hormone replacement therapy, skin diseases without systemic therapy and celiac disease which is fully controlled.
4. HIV-Ab, TP-Ab, HCV-Ab, HBsAg, HBeAg, HBeAb or HBcAb positive.
5. Any symptom, sign or laboratory examination abnormality suggesting acute or subacute infection (e.g. fever, cough, urinary irritation, skin infectious wound).
6. Female who are pregnant or cannot stop lactating.
7. Those who cannot communicate with medical staff due to mental illness or language disabilities.
8. Other unsuitable conditions that investigators believe unsuitable for the donation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Incidence of Adverse events (AEs) | up to 48 weeks
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Safety evaluation: Dose limited toxicity (DLTs) | up to 48 weeks
  The incidence, characteristic and severity of DLTs will be recorded and assessed.
Safety evaluation: Maximum-tolerated dose (MTD) | up to 48 weeks
  MTD or clinical recommended dose will be recorded and evaluated.

SECONDARY OUTCOMES:
Efficacy evaluation: Quality of life by ECOG score | up to 48 weeks
  The quality of life is assessed before and after the treatment by ECOG score .
Efficacy evaluation: Tumor markers | up to 48 weeks
  Tumor markers in peripheral blood will be tested and assessed (e. g. AFP, AFP-L3).
Efficacy evaluation: γδT cells in peripheral blood | up to 48 weeks
  Number and phenotype of γδT cells in peripheral blood will be assessed by flow cytometry.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing 302 Hospital of China, Beijing, Beijing Municipality
  - Beijing 302 hospital, Beijing